CLINICAL TRIAL: NCT06418230
Title: EXOME SEQUENCING IN MEDULLARY SPONGE KIDNEY
Acronym: EXOCARI
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23-5392
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Medulary Sponge Kidney
Keywords: exome; nephrolithiasis; medullary sponge kidney
MeSH Terms: conditions — Nephrolithiasis; Medullary Sponge Kidney

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 1 Urinary collection of the last 24 hours : Sodium, urea, creatinin, calcium, uric acid, oxalate, citrate, magnesium, albumin
  1 Urine sample : CBEU, UB, cristallury, Ca/creat
  1 Blood sample (20mL), including ionogram, albumin, creatinin, GFR (CKDEPI) (3mL) (3mL) ; PTH (4mL) ; 1-25 diOH Vit D (calcitriol) (4mL) ; 25OH Vit D (4mL)
  1 blood sample (4mL) : exome analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MEDULLARY SPONGE KIDNEY: medullary sponge kidney attending medical consultation

SUMMARY:
Medullary sponge kidney is a rare, underdiagnosed renal pathology, characterized by precalyceal dilatation of the renal tubes associated with active and recurrent stone disease with nephrocalcinosis, hypercalciuria and tubular dysfunction with, for example, acidification and urinary concentration defects.

The pathophysiology is poorly understood The prevalence and etiopathogenesis of the disease is not known Medullary sponge kidney is often characterized as a congenital pathology with delayed expression due to reported cases occurring in early childhood and associations with other congenital renal and extra-renal malformative pathologies, such as Wilms tumors, horseshoe kidney, contralateral renal hypoplasia, Beckwith-Wiedemann syndrome, Caroli disease, or congenital hepatic fibrosis, for example. However, no clear demonstration of the congenital nature has been established so far, and it is considered a sporadic disease.

However familial cases have been reported with an autosomal dominant mode.

The pathophysiology may involve disruptions in renal organogenesis, which depends on reciprocal inductive interactions necessary to coordinate nephrogenesis between the ureteric bud and the metanephric blastema during the 5th week of embryonic development. Some authors suggested that the GDNF and RET genes may be involved in the physiopathology of the disease.

For instance 12% of heterozygous patients for rare GDNF variants were identified in an Italian cohort of 57 medullary sponge kidney patients.

Other genes have been suggested to be involved in the pathophysiology based on reported cases, with no direct relationship demonstrated and their role remain putative Medullary sponge kidney disease is a debilitating condition, with the main symptoms being recurrent kidney stones and urinary infections.

Additional data are needed to determine the involvement of genetic anomalies in the pathophysiology of the condition.

The aim of the study is to describe the genetic variants identified with exome sequencing in medullary sponge kidney patients, in order to optimize management, especially for familial forms, and therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* medullary sponge kidney attending medical consultation
* consent signed
* affiliated to social insurance scheme

Exclusion Criteria:

* legal protection measure (guardianship, curatorship)
* Deprived of liberty by a judicial or administrative decision
* subject participating in another research including an exclusion period still in progress at inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The patients will be selected from the hospital Edouard Herriot nephrology and urology departments and frome from the hospital de la Conception nephrology and urology departments Around 80 Medullary sponge kidney patients are followed at these nephrology and urology departments
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Class 3, 4 and 5 variants detected at exome-sequencing | Baseline

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Edouard Herriot, Lyon
  - Hôpital de la Conception, Marseille